CLINICAL TRIAL: NCT07403682
Title: Comparison of M-TAPA and ESPB Blocks for Postoperative Analgesia After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: M-TAPA vs ESPB for Postoperative Analgesia After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCS-MTAPA-01
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain After Laparoscopic Cholecystectomy
Keywords: Laparoscopic cholecystectomy; M-TAPA block; Erector spinae plane block; Regional anesthesia; Postoperative analgesia; Opioid consumption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-TAPA Block (Experimental): An ultrasound-guided modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) performed bilaterally using local anesthetic for postoperative analgesia after laparoscopic cholecystectomy.
  Interventions: Procedure: Modifiye throcoabdominal nerve block through the perichondrial approach (M-TAPA)
- ESPB (Experimental): An ultrasound-guided erector spinae plane block (ESPB) performed using local anesthetic for postoperative analgesia after laparoscopic cholecystectomy.
  Interventions: Procedure: erector spinae plane block (ESPB)

INTERVENTIONS:
Procedure: Modifiye throcoabdominal nerve block through the perichondrial approach (M-TAPA) — An ultrasound-guided modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) performed bilaterally using local anesthetic for postoperative analgesia after laparoscopic cholecystectomy.
  Arms: M-TAPA Block
Procedure: erector spinae plane block (ESPB) — An ultrasound-guided erector spinae plane block (ESPB) performed using local anesthetic for postoperative analgesia after laparoscopic cholecystectomy.
  Arms: ESPB

SUMMARY:
Postoperative pain after laparoscopic cholecystectomy can negatively affect patient comfort, recovery, and opioid consumption. Regional abdominal wall blocks are commonly used as part of multimodal analgesia to improve postoperative pain control and reduce opioid-related side effects.

The modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) and the erector spinae plane block (ESPB) are two ultrasound-guided regional anesthesia techniques that have been shown to provide effective postoperative analgesia in abdominal surgery. However, comparative clinical data between these two techniques in laparoscopic cholecystectomy are limited.

This randomized, single-blind clinical trial aims to compare the postoperative analgesic effectiveness of M-TAPA and ESPB in adult patients undergoing elective laparoscopic cholecystectomy. Postoperative pain scores, opioid consumption, time to first analgesic requirement, and patient satisfaction will be evaluated.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, single-blind controlled clinical trial conducted in adult patients scheduled for elective laparoscopic cholecystectomy. The primary objective of the study is to compare the postoperative analgesic effectiveness of the modified thoracoabdominal nerve block through the perichondrial approach (M-TAPA) and the erector spinae plane block (ESPB).

Eligible patients aged 18 to 65 years with American Society of Anesthesiologists (ASA) physical status I-II will be randomly assigned in a 1:1 ratio to receive either M-TAPA or ESPB. Randomization will be performed using a computer-generated random number sequence, and allocation will be concealed in sealed, opaque envelopes to prevent selection bias.

All blocks will be performed under ultrasound guidance by experienced anesthesiologists using standard local anesthetic agents routinely applied in clinical practice. The study is designed as single-blind, with patients blinded to group allocation.

Postoperative pain intensity will be assessed using the visual analog scale (VAS) at 0, 1, 6, 12, and 24 hours after surgery. Additional outcome measures include total opioid consumption within the first 24 postoperative hours, time to first analgesic requirement, need for rescue analgesia, and patient satisfaction. Adverse events related to regional anesthesia techniques will be recorded.

The study follows the principles of the Declaration of Helsinki and Good Clinical Practice guidelines. Ethical approval has been obtained from the relevant Clinical Research Ethics Committee prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* ASA physical status I-III
* Scheduled for elective surgery under general anesthesia
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Refusal to participate
* Known allergy to local anesthetics
* Coagulation disorders or anticoagulant therapy
* Infection at the injection site
* Severe hepatic, renal, or cardiac disease
* Chronic opioid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption in the First 24 Hours | within the first 24 hours postoperatively
  Total cumulative opioid consumption within the first 24 hours after surgery, recorded as intravenous tramadol equivalent dose.

IPD SHARING:
Plan to Share IPD: No